CLINICAL TRIAL: NCT06440304
Title: Therapeutic Strategies for Carbapenem-Resistant Acinetobacter Baumannii Infections: Study Protocol
Brief Title: Therapeutic Options for CRAB
Acronym: TheraCRAB
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Ivan Šitum, MD, Principal invesigator, Clinical Hospital Centre Zagreb
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRAB01
Record Dates: First submitted 2024-05-21; First posted 2024-06-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Infections, Bacterial; Sepsis Bacterial
Keywords: Carbapenem-resistant Acinetobacter baumannii (CRAB); Intensive Care Unit (ICU) infections; Polymyxins (colistin); Combination antimicrobial therapy; Antimicrobial resistance mechanisms; Fosfomycin; Eravacyclin; Ampicillin/sulbactam
MeSH Terms: conditions — Bacterial Infections; Infections | interventions — Fosfomycin; Colistin; eravacycline; sultamicillin; Sulbactam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fosfomycin (Active Comparator): Upon the detection of a positive microbiological finding for A. baumannii, the Fosfomycin group will receive 8 grams of fosfomycin every 8 hours, along with an initial colistin bolus of 6 million IU, followed by 3 million IU every 8 hours. After the first day, the dosage will be adjusted based on kidney and liver function. This therapy will be administered for a total of 10 days.
  Interventions: Drug: Fosfomycin
- Ampicilin/sulbactam (Active Comparator): Upon the detection of a positive microbiological finding for A. baumannii, the Ampicilin/sulbactam group will receive an initial bolus dose of 2 grams of ampicillin and 1 gram of sulbactam, followed by a continuous infusion of 8 grams of ampicillin and 4 grams of sulbactam over 24 hours (maximum daily dose of 12 grams per day), along with a colistin bolus of 6 million IU, followed by 3 million IU every 8 hours. After the first day, the dosage will be adjusted based on kidney and liver function. This therapy will be administered for a total of 10 days.
  Interventions: Drug: ampicillin/sulbactam
- Eravacyclin (Active Comparator): Upon the detection of a positive microbiological finding for A. baumannii, the Eravacyclin group will receive eravacycline at a dose of 1 mg/kg every 12 hours for 60 minutes, along with a colistin bolus of 6 million IU, followed by 3 million IU every 8 hours. After the first day, the dosage will be adjusted based on kidney and liver function. This therapy will be administered for a total of 10 days.
  Interventions: Drug: Eravacycline

INTERVENTIONS:
Drug: Fosfomycin — Patients will be randomly divided according to a predetermined randomization table Upon arrival of a positive microbiological finding on A. baumannii, patient will be randomised to one of groups (Colistin with Unasyn OR Colistin with Xerava OR Colistin with Fosfomycin
  Other Names: Fosfomycin with Colistin
  Arms: Fosfomycin
Drug: Eravacycline — Patients will be randomly divided according to a predetermined randomization table Upon arrival of a positive microbiological finding on A. baumannii, patient will be randomised to one of groups (Colistin with Unasyn OR Colistin with Xerava OR Colistin with Fosfomycin
  Other Names: Eravacycline with Colistin
  Arms: Eravacyclin
Drug: ampicillin/sulbactam — Patients will be randomly divided according to a predetermined randomization table Upon arrival of a positive microbiological finding on A. baumannii, patient will be randomised to one of groups (Colistin with Unasyn OR Colistin with Xerava OR Colistin with Fosfomycin
  Other Names: Ampicilin/sulbactam with Colistin
  Arms: Ampicilin/sulbactam

SUMMARY:
CRAB infections in ICUs are on the rise, leading to higher morbidity, mortality, and healthcare costs due to resistance to most antibiotics, including carbapenems. The main resistance mechanisms include carbapenemases, efflux pumps, and changes in the bacterial cell wall.

Current treatments include polymyxins (Colistin, Polymyxin B), which are effective but can lead to resistance, aminoglycosides (Amikacin, Gentamicin), which are limited by resistance, and tetracyclines (Tigecycline, Eravacycline), which are effective against CRAB. Fosfomycin is effective in combination treatments, and combination therapy (e.g., colistin with sulbactam, fosfomycin, or eravacycline) can enhance outcomes.

Previous research shows promise for combination therapies, improving treatment efficacy and reducing mortality. New regimens are being studied to find optimal combinations. Individualized dosing is crucial, considering patient-specific factors like age, weight, and renal function. Adjustments depend on the infection site and comorbidities.

Strict infection control and antimicrobial stewardship programs (ASPs) are essential. ASPs focus on optimizing antibiotic use and reducing resistance through education and surveillance. Future directions include continued research for new drugs or combinations and strategies to overcome resistance and improve treatment efficacy.

Study goals include achieving negative samples after 10 days of therapy, 30-day survival, discharge rates, reduced SOFA scores, and improved clinical and radiological findings. A randomized study will compare colistin combined with fosfomycin, ampicillin/sulbactam, and eravacycline.

In summary, treating CRAB infections is complex, requiring combination therapy, individualized dosing, and strict infection control measures.

DETAILED DESCRIPTION:
The primary goal will be to negativize positive samples (surveillance or diagnostic) after 10 days of therapy. In addition to the control samples with the same name, samples will be taken on the 4th, 7th, and 10th day after starting treatment.

The secondary objectives will include 30-day survival, discharge from the ICU, discharge from the hospital, reduction in SOFA score, rate of reinfection, and frequency of complications (deterioration of renal function). Reduction of CRP, PCT, and leukocytes, improvement of the clinical picture, improvement of radiological findings (such as X-ray of the lungs), and reduction of elevated body temperature will also be included.

Patients who require treatment in the ICU with a positive sample (surveillance or diagnostic) for A. baumannii, with clinical signs of infection (temperature >38.5, CPR >50, L >10000) (in which no infection can be explained by another cause) will be included.

Three groups will be formed:

1. colistin + fosfomycin
2. colistin + ampicilin/sulbactam
3. colistin + eravacyclin

The outcomes will include a negative sample, length of stay in the ICU, length of stay in the hospital, and reduction of SOFA score.

The hypothesis will be that the combination of fosfomycin with colistin and eravacyclin with colistin will lead to faster negative samples than the combination of ampicillin/sulbactam with colistin in intensive care unit patients diagnosed with carbapenem-resistant A. baumannii.

After obtaining approval from the ethics committee of KBC Zagreb, this study will be conducted at the UHC Zagreb, Department of Anesthesiology and ICU. Patients will be randomly divided according to a predetermined randomization table.

Upon arrival of a positive microbiological finding on A. baumannii, the Fosfomycin group will receive fosfomycin 8 g every 8 h, together with a colistin bolus of 6 million IJ, followed by 3 million IJ every 8 h. After the first day, the dose will be adjusted according to kidney and liver function. Therapy will be administered for 10 days.

Upon arrival of a positive microbiological finding on A. baumannii, the Ampicilin/sulbactam group will receive a bolus dose of ampicillin/sulbactam 2 g + 1 g and a continuous infusion of 8 g + 4 g over 24 h together (maximum daily dose 12 g/day) with a colistin bolus of 6 million IJ, followed by 3 million IJ every 8 h. After the first day, the dose will be adjusted according to kidney and liver function. Therapy will be performed for 10 days.

Upon arrival of a positive microbiological finding for A. baumannii, the Eravacyclin group will receive eravacycline at a dose of 1 mg/kg every 12 h for 60 min together with a colistin bolus of 6 million IU, and then 3 million IU every 8 h. After the first day, the dose will be adjusted according to kidney and liver function. Therapy will be administered for 10 days.

After the first positive microbiological finding for A. baumannii, the test will be repeated on the 4th, 7th, and 10th days from the start of therapy. The Charlson Comorbidity Index will be calculated for each patient upon inclusion in the study. The SOFA score will be calculated daily for each patient over 10 days.

Patient data from a hospital information system will be used in this study. Demographic data, comorbidities, habits (alcohol and cigarettes), Charlson comorbidity index, SOFA score, allergies, and the type of positive sample will be recorded. The Charlson Comorbidity Index will be calculated for each patient upon inclusion in the study. The SOFA score will be calculated daily for each patient over 10 days. Patients will be included in the study after the arrival of a microbiological test positive for A. baumannii. A routine antimicrobial susceptibility test will be performed when the microbiological findings are positive for A. baumannii. The sensitivity of all A. baumannii strains included in the study, regardless of the group to which they belonged (fosfomycin, ampicilin/sulbactam, and eravacyclin), will be determined during the microbiological analysis of all A. baumannii strains included in the study. After the first positive microbiological finding for A. baumannii, the test will be repeated on the 3th, 7th, and 10th days from the start of therapy. For each patient included in the study, inflammatory parameters (leukocytes, CRP, procalcitonin) and the number of days and discharge from the ICU and hospital as well as 30-day mortality and cause of death, complications (AKI and ALF), and reinfection will be monitored.

For a test power of 80% and the use of an independent t-test for the primary objective and a chi-square test for the secondary objective with a statistical significance of 0.05, it will be necessary to include 108 patients, divided into three groups, with 36 subjects per group. The test for power calculation will be conducted using G Power Version 3.1.9.6. The results will be processed using IBM SPSS Statistics v27.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients (abdominal, vascular, and polytraumatized patients)
* Older than 18 years
* Require postoperative treatment in the ICU
* A positive sample (surveillance or diagnostic) for A. baumannii with signs of systemic infection

Infection will be defined as a diagnostic microbiologically positive sample for A. baumannii and a surveillance microbiologically positive sample for A. baumannii with signs of systemic infection (elevated CRP, leukocytes, and body temperature).

Colonization will be defined as a positive surveillance microbiological sample for A. baumannii in the absence of signs of systemic infection (normal CRP, leukocytes, and body temperature).

Exclusion Criteria:

* Allergy to the study medications
* Positive surveillance swabs for A. baumannii without signs of systemic infection
* Positive findings (surveillance or diagnostic) for carbapenem-sensitive A. baumannii
* Refusal to participate in the research

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Negativisation | 10 days
  Rate of negativisation of (surveillance or diagnostic) microbiological sample;

SECONDARY OUTCOMES:
Length of stay in ICU | 90 days
  Days spent in ICU total after randomisation
Length of stay in hospital | 90 days
  Days spent in hospital total after randomisation
Reduction of Sequential Organ Failure Assessment (SOFA) score | 10 days
  Change in initial SOFA score from randomisation day, from 0 points to 24

OTHER OUTCOMES:
30 day Survival | 30 day
  patients survived 30 days after randomisation
Reduction of inflamatory parameters | 10 days
  Reduction of parameters of inflamation (L,CRP, PCT)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Šitum, Principal Investigator — UHC Zagreb
Locations (1):
- University Hospital Centre Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Šitum I, Mamić G, Džaja N, Hrvoić L, Lovrić D, Siroglavić M, et al. Upala pluća povezana s mehaničkom ventilacijom uzrokovana bakterijom Acinetobacter baumannii u razdoblju pandemije COVID-19. Medicina Fluminensis : Medicina Fluminensis [Internet]. 2023 Jun 1 [cited 2024 Apr 30];59(2):139-48. Available from: http://hrcak.srce.hr/medicinamedicinafluminensis
- [Background] Carbapenem-resistant Acinetobacter baumannii (CRAB): An urgent public health threat in United States healthcare facilities | A.R. & Patient Safety Portal [Internet]. [cited 2024 May 2]. Available from: https://arpsp.cdc.gov/story/cra-urgent-public-health-threat
- [Background] Shields RK, Paterson DL, Tamma PD. Navigating Available Treatment Options for Carbapenem-Resistant Acinetobacter baumannii-calcoaceticus Complex Infections. Clin Infect Dis. 2023 May 1;76(Suppl 2):S179-S193. doi: 10.1093/cid/ciad094. PMID 37125467
- [Background] Isler B, Doi Y, Bonomo RA, Paterson DL. New Treatment Options against Carbapenem-Resistant Acinetobacter baumannii Infections. Antimicrob Agents Chemother. 2018 Dec 21;63(1):e01110-18. doi: 10.1128/AAC.01110-18. Print 2019 Jan. PMID 30323035
- [Background] Viehman JA, Nguyen MH, Doi Y. Treatment options for carbapenem-resistant and extensively drug-resistant Acinetobacter baumannii infections. Drugs. 2014 Aug;74(12):1315-33. doi: 10.1007/s40265-014-0267-8. PMID 25091170
- [Background] Dalfino L, Stufano M, Bavaro DF, Diella L, Belati A, Stolfa S, Romanelli F, Ronga L, Di Mussi R, Murgolo F, Loconsole D, Chironna M, Mosca A, Montagna MT, Saracino A, Grasso S. Effectiveness of First-Line Therapy with Old and Novel Antibiotics in Ventilator-Associated Pneumonia Caused by Carbapenem-Resistant Acinetobacter baumannii: A Real Life, Prospective, Observational, Single-Center Study. Antibiotics (Basel). 2023 Jun 14;12(6):1048. doi: 10.3390/antibiotics12061048. PMID 37370367
- [Background] Paul M, Carrara E, Retamar P, Tangden T, Bitterman R, Bonomo RA, de Waele J, Daikos GL, Akova M, Harbarth S, Pulcini C, Garnacho-Montero J, Seme K, Tumbarello M, Lindemann PC, Gandra S, Yu Y, Bassetti M, Mouton JW, Tacconelli E, Rodriguez-Bano J. European Society of Clinical Microbiology and Infectious Diseases (ESCMID) guidelines for the treatment of infections caused by multidrug-resistant Gram-negative bacilli (endorsed by European society of intensive care medicine). Clin Microbiol Infect. 2022 Apr;28(4):521-547. doi: 10.1016/j.cmi.2021.11.025. Epub 2021 Dec 16. PMID 34923128
- [Background] Rodrigues RD, Garcia RCL, Bittencourt GA, Waichel VB, Garcia ECL, Rigatto MH. Antimicrobial Therapy Duration for Bloodstream Infections Caused by Pseudomonas aeruginosa or Acinetobacter baumannii-calcoaceticus complex: A Retrospective Cohort Study. Antibiotics (Basel). 2023 Mar 8;12(3):538. doi: 10.3390/antibiotics12030538. PMID 36978405
- [Background] Reina R, Leon-Moya C, Garnacho-Montero J. Treatment of Acinetobacter baumannii severe infections. Med Intensiva (Engl Ed). 2022 Dec;46(12):700-710. doi: 10.1016/j.medine.2022.08.007. Epub 2022 Oct 19. PMID 36272902
- [Background] Acinetobacter in Healthcare Settings | HAI | CDC [Internet]. [cited 2024 Apr 30]. Available from: https://www.cdc.gov/hai/organisms/acinetobacter.html
- [Background] Nartey YA, Donkor AB, Siaw ADJ, Ekor OE, Jimah BB. Carbapenem-Resistant Acinetobacter baumannii Bloodstream Infection in a Ghanaian Patient with Unilateral Diaphragmatic Eventration and HIV Type 1 Infection. Case Rep Infect Dis. 2023 Oct 12;2023:9930291. doi: 10.1155/2023/9930291. eCollection 2023. PMID 37867582
- [Background] Kim SH, Wi YM, Peck KR. Clinical Effectiveness of Tetracycline-Class Agents Based Regimens in Patients With Carbapenem-Resistant Acinetobacter baumannii Bacteremia: A Single-Center Retrospective Cohort Study. J Korean Med Sci. 2023 Aug 28;38(34):e263. doi: 10.3346/jkms.2023.38.e263. PMID 37644679
- [Background] Jung SY, Lee SH, Lee SY, Yang S, Noh H, Chung EK, Lee JI. Antimicrobials for the treatment of drug-resistant Acinetobacter baumannii pneumonia in critically ill patients: a systemic review and Bayesian network meta-analysis. Crit Care. 2017 Dec 20;21(1):319. doi: 10.1186/s13054-017-1916-6. PMID 29262831
- [Background] Pogue JM, Zhou Y, Kanakamedala H, Cai B. Burden of illness in carbapenem-resistant Acinetobacter baumannii infections in US hospitals between 2014 and 2019. BMC Infect Dis. 2022 Jan 6;22(1):36. doi: 10.1186/s12879-021-07024-4. PMID 34991499
- [Background] Seok H, Choi WS, Lee S, Moon C, Park DW, Song JY, Cheong HJ, Kim J, Kim JY, Park MN, Kim YR, Lee HJ, Kim B, Pai H, Jo YM, Kim JH, Sohn JW. What is the optimal antibiotic treatment strategy for carbapenem-resistant Acinetobacter baumannii (CRAB)? A multicentre study in Korea. J Glob Antimicrob Resist. 2021 Mar;24:429-439. doi: 10.1016/j.jgar.2021.01.018. Epub 2021 Feb 8. PMID 33571708
- [Background] Gatti M, Viaggi B, Rossolini GM, Pea F, Viale P. An Evidence-Based Multidisciplinary Approach Focused on Creating Algorithms for Targeted Therapy of Infection-Related Ventilator-Associated Complications (IVACs) Caused by Pseudomonas aeruginosa and Acinetobacter baumannii in Critically Ill Adult Patients. Antibiotics (Basel). 2021 Dec 28;11(1):33. doi: 10.3390/antibiotics11010033. PMID 35052910
- [Background] Ozger HS, Cuhadar T, Yildiz SS, Demirbas Gulmez Z, Dizbay M, Guzel Tunccan O, Kalkanci A, Simsek H, Unaldi O. In vitro activity of eravacycline in combination with colistin against carbapenem-resistant A. baumannii isolates. J Antibiot (Tokyo). 2019 Aug;72(8):600-604. doi: 10.1038/s41429-019-0188-6. Epub 2019 Apr 26. PMID 31028352
- [Background] Abdallah M, Olafisoye O, Cortes C, Urban C, Landman D, Quale J. Activity of eravacycline against Enterobacteriaceae and Acinetobacter baumannii, including multidrug-resistant isolates, from New York City. Antimicrob Agents Chemother. 2015 Mar;59(3):1802-5. doi: 10.1128/AAC.04809-14. Epub 2014 Dec 22. PMID 25534744
- [Background] Monogue ML, Thabit AK, Hamada Y, Nicolau DP. Antibacterial Efficacy of Eravacycline In Vivo against Gram-Positive and Gram-Negative Organisms. Antimicrob Agents Chemother. 2016 Jul 22;60(8):5001-5. doi: 10.1128/AAC.00366-16. Print 2016 Aug. PMID 27353265
- [Background] Zhanel GG, Baxter MR, Adam HJ, Sutcliffe J, Karlowsky JA. In vitro activity of eravacycline against 2213 Gram-negative and 2424 Gram-positive bacterial pathogens isolated in Canadian hospital laboratories: CANWARD surveillance study 2014-2015. Diagn Microbiol Infect Dis. 2018 May;91(1):55-62. doi: 10.1016/j.diagmicrobio.2017.12.013. Epub 2017 Dec 22. PMID 29338931
- [Background] Ni W, Shao X, Di X, Cui J, Wang R, Liu Y. In vitro synergy of polymyxins with other antibiotics for Acinetobacter baumannii: a systematic review and meta-analysis. Int J Antimicrob Agents. 2015 Jan;45(1):8-18. doi: 10.1016/j.ijantimicag.2014.10.002. Epub 2014 Oct 24. PMID 25465524
- [Background] Grabein B, Graninger W, Rodriguez Bano J, Dinh A, Liesenfeld DB. Intravenous fosfomycin-back to the future. Systematic review and meta-analysis of the clinical literature. Clin Microbiol Infect. 2017 Jun;23(6):363-372. doi: 10.1016/j.cmi.2016.12.005. Epub 2016 Dec 9. PMID 27956267
- [Background] Assimakopoulos SF, Karamouzos V, Eleftheriotis G, Lagadinou M, Bartzavali C, Kolonitsiou F, Paliogianni F, Fligou F, Marangos M. Efficacy of Fosfomycin-Containing Regimens for Treatment of Bacteremia Due to Pan-Drug Resistant Acinetobacter baumannii in Critically Ill Patients: A Case Series Study. Pathogens. 2023 Feb 9;12(2):286. doi: 10.3390/pathogens12020286. PMID 36839558
- [Background] Nwabor OF, Terbtothakun P, Voravuthikunchai SP, Chusri S. Evaluation of the Synergistic Antibacterial Effects of Fosfomycin in Combination with Selected Antibiotics against Carbapenem-Resistant Acinetobacter baumannii. Pharmaceuticals (Basel). 2021 Feb 25;14(3):185. doi: 10.3390/ph14030185. PMID 33668905
- [Background] Mohd Sazlly Lim S, Heffernan A, Naicker S, Wallis S, Roberts JA, Sime FB. Evaluation of Fosfomycin-Sulbactam Combination Therapy against Carbapenem-Resistant Acinetobacter baumannii Isolates in a Hollow-Fibre Infection Model. Antibiotics (Basel). 2022 Nov 9;11(11):1578. doi: 10.3390/antibiotics11111578. PMID 36358238
- [Background] Warrier AR, Sneha R, Wilson A, Prakash S. 654. Clinical efficacy and safety of high dose Ampicillin sulbactam among patients with CRAB infections: A case series. Open Forum Infect Dis [Internet]. 2022 Dec 15 [cited 2024 Apr 30];9(Supplement_2). Available from: https://dx.doi.org/10.1093/ofid/ofac492.706
- [Background] Saelim W, Changpradub D, Thunyaharn S, Juntanawiwat P, Nulsopapon P, Santimaleeworagun W. Colistin plus Sulbactam or Fosfomycin against Carbapenem-Resistant Acinetobacter baumannii: Improved Efficacy or Decreased Risk of Nephrotoxicity? Infect Chemother. 2021 Mar;53(1):128-140. doi: 10.3947/ic.2021.0007. PMID 34409786
- [Background] Cunha BA. Optimal therapy for multidrug-resistant Acinetobacter baumannii. Emerg Infect Dis. 2010 Jan;16(1):170; author reply 170-1. doi: 10.3201/eid1601.091467. No abstract available. PMID 20031080
- [Background] Bartal C, Rolston KVI, Nesher L. Carbapenem-resistant Acinetobacter baumannii: Colonization, Infection and Current Treatment Options. Infect Dis Ther. 2022 Apr;11(2):683-694. doi: 10.1007/s40121-022-00597-w. Epub 2022 Feb 17. PMID 35175509